CLINICAL TRIAL: NCT01829009
Title: Resistance Exercise Effect on Physical Performance and Functional Status in Sarcopenic Older Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial issues
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, José Alberto Ávila Funes, PhD, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GER-887-13/14-1
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Elderly; Women; Resistance; Exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Recommendations Group (No Intervention): General information about sarcopenia will be provided to the participants, as well as general recommendations of healthy habits. We will contact the participants weekly by phone to answer questions about sarcopenia, and remind them of their next appointment and about adverse events occured during this period of time. The frequent contact with the participants has also the purpose to prevent losses or rejections for future evaluations
- Resistance Exercise Group (Experimental): An individualized resistance exercise program wil be applied twice a week by an expert physiotherapist. Every 2 weeks, intensity will be reassessed by the same physiotherapist. Weekly, participants will be asked about incidents such as the occurrence of falls or hospitalizations during this study period.
  Physical performance and functional status will be assessed by the blind investigator at weeks 6,12 and 24
  Interventions: Other: Resistance Exercise Group

INTERVENTIONS:
Other: Resistance Exercise Group — An individualized resistance exercise program wil be applied twice a week by an expert physiotherapist. Every 2 weeks, intensity will be reassessed by the same physiotherapist. Weekly, participants will be asked about incidents such as the occurrence of falls or hospitalizations during this study period.
  Physical performance and functional status will be assessed by the blind investigator at weeks 6,12 and 24
  Arms: Resistance Exercise Group

SUMMARY:
Aging is characterized by a progressive loss of multiple physical and cognitive abilities. From these changes, the most important one is the loss of muscle mass, which has been called "sarcopenia". Resistance exercise is a therapeutic approach for sarcopenia, nevertheless there is no universal consensus. Therefore, this research is interested in determining the effect of a resistance exercise program on physical performance and/or functional status in sarcopenic older women. The main study hypothesis is that a program of resistance exercise will improve physical performance and functional status in sarcopenic older women compared against general recommendations.

This is a single-blind, controlled clinical trial, including women> 70 years, living in the community with sarcopenia. Those who agree to participate, will be randomly assigned to one of the following groups:

1. Resistance Exercise Group
2. General Recommendations Group (control) The study will last 24 weeks, with 4 measurements performed at baseline, week 6, 12 and 24. Multilevel models (random effects) will be constructed for the comparison between the two groups. Tests will be conducted with a P=0.05 and confidence intervals at 95%. This protocol has been approved by the local ethics committee.

DETAILED DESCRIPTION:
Study withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Body mass composition by BIA with skeletal muscle mass <6.76kg/m2
* Speed gait of <0.8m/sec
* Handgrip strength (adjusted for BMI) less than 20kg

Exclusion Criteria:

* Current diagnosis of malnutrition (BMI <19kg/m2)
* Decompensated heart failure (NYHA III or IV)
* Hemiplegia or hemiparesis due to cerebral vascular disease
* Exacerbation of chronic obstructive pulmonary disease
* Dementia (any type, moderate or severe stage)
* Uncontrolled diabetes mellitus (glycosylated hemoglobin >8%)
* Severe pain in hips, knees or ankles
* Fracture of lower limb in the last 6 months
* Myocardial infarction within the past 6 months
* Severe hypertension (SBP > 180mmHg or DBP > 110 mmHg)
* Orthostatic hypotension

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Improvement in gait speed and functional status in sarcopenic older women | improvement in gait speed and functional status in sarcopenic older women in weeks 6,12 and 24

SECONDARY OUTCOMES:
Increase in muscle mass in sarcopenic older women | Increase in muscle mass in sarcopenic older women in week 24

CONTACTS AND LOCATIONS:
Overall Officials: JOSE ALBERTO AVILA FUNES, MD PhD, Principal Investigator — GERIATRICS CHIEF DEPARTMENT
Locations (1):
- National Institue of Medical Sciences and Nutrition Salvador Zubirán, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Rosenberg IH. Sarcopenia: origins and clinical relevance. J Nutr. 1997 May;127(5 Suppl):990S-991S. doi: 10.1093/jn/127.5.990S. PMID 9164280
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Yarasheski KE, Zachwieja JJ, Bier DM. Acute effects of resistance exercise on muscle protein synthesis rate in young and elderly men and women. Am J Physiol. 1993 Aug;265(2 Pt 1):E210-4. doi: 10.1152/ajpendo.1993.265.2.E210. PMID 8368290
- [Background] Baumgartner RN, Koehler KM, Gallagher D, Romero L, Heymsfield SB, Ross RR, Garry PJ, Lindeman RD. Epidemiology of sarcopenia among the elderly in New Mexico. Am J Epidemiol. 1998 Apr 15;147(8):755-63. doi: 10.1093/oxfordjournals.aje.a009520. PMID 9554417
- [Background] Visser M, Kritchevsky SB, Goodpaster BH, Newman AB, Nevitt M, Stamm E, Harris TB. Leg muscle mass and composition in relation to lower extremity performance in men and women aged 70 to 79: the health, aging and body composition study. J Am Geriatr Soc. 2002 May;50(5):897-904. doi: 10.1046/j.1532-5415.2002.50217.x. PMID 12028178
- [Background] Visser M, Harris TB, Langlois J, Hannan MT, Roubenoff R, Felson DT, Wilson PW, Kiel DP. Body fat and skeletal muscle mass in relation to physical disability in very old men and women of the Framingham Heart Study. J Gerontol A Biol Sci Med Sci. 1998 May;53(3):M214-21. doi: 10.1093/gerona/53a.3.m214. PMID 9597054
- [Background] Janssen I, Heymsfield SB, Baumgartner RN, Ross R. Estimation of skeletal muscle mass by bioelectrical impedance analysis. J Appl Physiol (1985). 2000 Aug;89(2):465-71. doi: 10.1152/jappl.2000.89.2.465. PMID 10926627
- [Background] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177
- [Background] Kim HK, Suzuki T, Saito K, Yoshida H, Kobayashi H, Kato H, Katayama M. Effects of exercise and amino acid supplementation on body composition and physical function in community-dwelling elderly Japanese sarcopenic women: a randomized controlled trial. J Am Geriatr Soc. 2012 Jan;60(1):16-23. doi: 10.1111/j.1532-5415.2011.03776.x. Epub 2011 Dec 5. PMID 22142410
- [Background] Velazquez MC, Irigoyen ME. Sarcopenia: Una entidad de relevancia clínica actual. Rev Cien Clin 2011;12(1):22-33
- [Background] Latham NK, Bennett DA, Stretton CM, Anderson CS. Systematic review of progressive resistance strength training in older adults. J Gerontol A Biol Sci Med Sci. 2004 Jan;59(1):48-61. doi: 10.1093/gerona/59.1.m48. PMID 14718486